CLINICAL TRIAL: NCT04434261
Title: Oncological Surgery in Times of COVID-19: Effectiveness of Preoperative Screening for Sars-Cov-2
Acronym: ASTANA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto Brasileiro de Controle do Cancer (Other)
Responsible Party: Sponsor
Other Study IDs: 33467320.0.0000.0072
Record Dates: First submitted 2020-06-15; First posted 2020-06-16 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: SARS-CoV-2; Oncology; Surgery
Keywords: SARS-CoV-2; Surgical Oncology; PT-PCR Screening Test
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients tested for SARS-CoV-2: Patients who underwent the preoperative screening program for SARS-CoV-2
  Interventions: Diagnostic Test: PT-PCR test for SARS-CoV-2

INTERVENTIONS:
Diagnostic Test: PT-PCR test for SARS-CoV-2 — Screening test for the diagnosis of SARS-CoV-2 in asymptomatic patients

SUMMARY:
To evaluate the incidence of patients with a positive test for SARS-CoV-2, performed in the preoperative screening for patients treated at the institution

DETAILED DESCRIPTION:
Cohort, prospective, observational study to evaluate the incidence of asymptomatic patients with a positive SARS-CoV-2 test detected in the preoperative screening program of the institution.

ELIGIBILITY:
Inclusion Criteria:

* Patients with elective surgery scheduled at the IBCC, including those diagnosed with any type of cancer;
* Patients who will undergo the screening test for SARS-COV-2 by RT-PCR (nasal swab), according to the guidelines and protocol of the hospital

Exclusion Criteria:

* Urgent or emergency surgery;
* Screening test for SARS-COV-2 not performed
* Incomplete data in the institutional database

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with scheduled elective surgery, including all types of cancer
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-05-11 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of patients with a positive test for SARS-CoV-2, detected in the preoperative screening program | May- December 2020
  Describe the incidence of patients with a positive test for SARS-CoV-2, detected in the preoperative screening program in our center

SECONDARY OUTCOMES:
Incidence of SARS-CoV-2 infection in the postoperative period in patients with negative screening test; | Up to 30 days
  Describe the incidence of SARS-CoV-2 infection in the postoperative period in patients with negative screening test.
Postoperative complications | Up to 30 days
  Postoperative complications will be recorded, according to the Clavien-Dindo classification.
Mortality | 30 days
  To evaluate the risk of all-cause mortality
Delay in the cancer treatment | May 2020- March 2021
  Assess the impact of delayed cancer treatment

CONTACTS AND LOCATIONS:
Overall Officials: Andre Lopes, MD, Principal Investigator — Instituto Brasileiro de Controle do Cancer
Locations (1):
- Instituto Brasileiro de Controle do Cancer - IBCC, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available in a scientific publication
Access Criteria: There are no sharing Access Criteria

REFERENCES:
- [Background] Shinde RS, Naik MD, Shinde SR, Bhandare MS, Chaudhari VA, Shrikhande SV, Dcruz AK. To Do or Not to Do?-A Review of Cancer Surgery Triage Guidelines in COVID-19 Pandemic. Indian J Surg Oncol. 2020 Jun;11(2):175-181. doi: 10.1007/s13193-020-01086-7. Epub 2020 May 11. PMID 32395064
- [Background] Liang W, Guan W, Chen R, Wang W, Li J, Xu K, Li C, Ai Q, Lu W, Liang H, Li S, He J. Cancer patients in SARS-CoV-2 infection: a nationwide analysis in China. Lancet Oncol. 2020 Mar;21(3):335-337. doi: 10.1016/S1470-2045(20)30096-6. Epub 2020 Feb 14. No abstract available. PMID 32066541
- [Background] Romanzi A, Galletti M, Macchi L, Putorti A, Rossi F, Scolaro R, Vannelli A. Awake laparotomy: is locoregional anesthesia a functional option for major abdominal surgeries in the COVID-19 era? Eur Rev Med Pharmacol Sci. 2020 May;24(9):5162-5166. doi: 10.26355/eurrev_202005_21211. PMID 32432781
- [Background] Wang H, Zhang L. Risk of COVID-19 for patients with cancer. Lancet Oncol. 2020 Apr;21(4):e181. doi: 10.1016/S1470-2045(20)30149-2. Epub 2020 Mar 3. No abstract available. PMID 32142621
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Dai M, Liu D, Liu M, Zhou F, Li G, Chen Z, Zhang Z, You H, Wu M, Zheng Q, Xiong Y, Xiong H, Wang C, Chen C, Xiong F, Zhang Y, Peng Y, Ge S, Zhen B, Yu T, Wang L, Wang H, Liu Y, Chen Y, Mei J, Gao X, Li Z, Gan L, He C, Li Z, Shi Y, Qi Y, Yang J, Tenen DG, Chai L, Mucci LA, Santillana M, Cai H. Patients with Cancer Appear More Vulnerable to SARS-CoV-2: A Multicenter Study during the COVID-19 Outbreak. Cancer Discov. 2020 Jun;10(6):783-791. doi: 10.1158/2159-8290.CD-20-0422. Epub 2020 Apr 28. PMID 32345594
- [Background] Tan KK, Moran BJ, Solomon MJ. Avoiding collateral mortality in a pandemic - time to change our mindset in surgical oncology. Nat Rev Clin Oncol. 2020 Jul;17(7):383-385. doi: 10.1038/s41571-020-0383-1. PMID 32372035
- [Background] Tuech JJ, Gangloff A, Di Fiore F, Michel P, Brigand C, Slim K, Pocard M, Schwarz L. Strategy for the practice of digestive and oncological surgery during the Covid-19 epidemic. J Visc Surg. 2020 Jun;157(3S1):S7-S12. doi: 10.1016/j.jviscsurg.2020.03.008. Epub 2020 Mar 31. PMID 32249098
- [Background] Schrag D, Hershman DL, Basch E. Oncology Practice During the COVID-19 Pandemic. JAMA. 2020 May 26;323(20):2005-2006. doi: 10.1001/jama.2020.6236. No abstract available. PMID 32282023
- [Background] Bourget-Murray J, Heard BJ, Bansal R, Johnson AS, Powell J. Postoperative fever in the time of COVID-19. Can J Surg. 2020 May 8;63(3):E231-E232. doi: 10.1503/cjs.004720. PMID 32386473
- [Background] Bartlett DL, Howe JR, Chang G, Crago A, Hogg M, Karakousis G, Levine E, Maker A, Mamounas E, McGuire K, Merchant N, Shibata D, Sohn V, Solorzano C, Turaga K, White R, Yang A, Yoon S; Society of Surgical Oncology. Management of Cancer Surgery Cases During the COVID-19 Pandemic: Considerations. Ann Surg Oncol. 2020 Jun;27(6):1717-1720. doi: 10.1245/s10434-020-08461-2. Epub 2020 Apr 8. No abstract available. PMID 32270420
- [Background] Tilmans G, Chenevas-Paule Q, Muller X, Breton A, Mohkam K, Ducerf C, Mabrut JY, Lesurtel M. Surgical outcomes after systematic preoperative severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) screening. Surgery. 2020 Aug;168(2):209-211. doi: 10.1016/j.surg.2020.05.006. Epub 2020 May 18. No abstract available. PMID 32425247
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] COVIDSurg Collaborative. Mortality and pulmonary complications in patients undergoing surgery with perioperative SARS-CoV-2 infection: an international cohort study. Lancet. 2020 Jul 4;396(10243):27-38. doi: 10.1016/S0140-6736(20)31182-X. Epub 2020 May 29. PMID 32479829
- [Background] Peak CM, Kahn R, Grad YH, Childs LM, Li R, Lipsitch M, Buckee CO. Individual quarantine versus active monitoring of contacts for the mitigation of COVID-19: a modelling study. Lancet Infect Dis. 2020 Sep;20(9):1025-1033. doi: 10.1016/S1473-3099(20)30361-3. Epub 2020 May 20. PMID 32445710
- [Background] Ganesh Kumar N, Drolet BC. COVID-19 - Implications on and of Surgical Practices: Where Do We Draw the Line? Ann Surg. 2020 Aug;272(2):e45-e46. doi: 10.1097/SLA.0000000000004009. No abstract available. PMID 32675491